CLINICAL TRIAL: NCT05054335
Title: CPRIT: Optimizing Surgical and Rehabilitation Treatment of Pelvic Sarcomas Using Computational Models
Brief Title: Patient-Specific Computational Walking Models in Improving Surgical and Rehabilitation Treatment in Patients With Pelvic Sarcomas
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-0216; NCI-2019-00862 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0216 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-03-07; First posted 2021-09-23 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Pelvic Sarcoma
MeSH Terms: interventions — X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supportive care (walking function test, X-ray) (Experimental): Patients undergo walking function assessment using optical motion capture and bi-plane dynamic X-ray imaging pre- and post-hemipelvectomy.
  Interventions: Other: Functional Assessment; Procedure: X-Ray Imaging
- Retrospective Group (No Intervention): 1. Acquisition of pre- and post-operative MRI data of the pelvic region (when available) collected previously as part of standard clinical care
  2. Acquisition of pre-operative CT data of the pelvic region (when available) collected previously as part of standard clinical care
  3. Acquisition of Physical Therapy Assessment data collected previously by a physical therapist and/or physical therapist assistant under protocol PA12-1046

INTERVENTIONS:
Other: Functional Assessment — Undergo walking function assessment with optical motion capture
  Arms: Supportive care (walking function test, X-ray)
Procedure: X-Ray Imaging — Undergo bi-plane dynamic X-ray imaging
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Radiography; Static X-Ray; X-Ray
  Arms: Supportive care (walking function test, X-ray)

SUMMARY:
This trial studies the development of patient-specific computational walking models to improve the surgical planning and rehabilitation treatment of patients with pelvic sarcomas. Every pelvis and pelvic sarcoma are different, and the orthopedic oncologist faces significant challenges when removing a tumor from the complex anatomy of the pelvis. These challenges make it difficult to achieve excellent oncological and functional outcomes together. Computational walking models may be used to predict the best combination of surgical methods and how to implement them to maximize each patient's post-surgery walking function.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To develop patient-specific computational walking models to predict the optimal combination of pelvic sarcoma surgical and rehabilitation decisions that will maximize each patient's post-surgery walking function.

II. To collect experimental movement and imaging data prospectively and retrospectively from individuals who have already received, or are going to receive, a type I or type II hemipelvectomy.

III. To use the data to develop computational modeling and simulation methodologies that can predict an individual patient's post-surgery walking function given pre-surgery movement and imaging data and the surgical decisions made by the surgeon.

OUTLINE:

Patients undergo walking function assessment using optical motion capture and bi-plane dynamic X-ray imaging pre- and post-hemipelvectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have received or are scheduled to receive an internal hemipelvectomy with or without reconstruction at UT MD Anderson Cancer Center.
2. Patients who are 18 years of age and older

Exclusion Criteria:

1. Patients who have undergone an external (hindquarter amputated), or an isolated type III internal hemipelvectomy.
2. Previous surgery or significant injury to either hip (prospective patients only)
3. Relevant surgery, procedure, injury, or condition in the last two years which may affect hip pain or general movement patterns on either side (prospective patients only)
4. Pregnant women or women nursing an infant
5. Persons with a pacemaker, hearing aid, aneurysm clips or artificial heart valves, and other forms of loose metal implants will be excluded from the study as assessed by a pre-MRI questionnaire administered by the MRI technician at the time of the scan.
6. Radiological exclusion criteria (assessed after MR scan is conducted on the first visit, prior to DSX/CT radiation exposure): evidence on preliminary MRI of fracture, slipped capital femoral epiphysis (SCFE), masses, lesions, or other anomalies not consistent with an FAI diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2019-06-20 (Actual); Primary Completion 2027-12-21 (Estimated); Study Completion 2027-12-21 (Estimated)

PRIMARY OUTCOMES:
To establish the patient-specific computational models to inform surgical decisions and design custom implants that maximize post-surgery function. | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Valerae O Lewis, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org